CLINICAL TRIAL: NCT02902458
Title: Psychological Intervention modifiEs Outcome of Patients With implAntable Cardioverter dEfibrillator: The PEACE Study
Acronym: PEACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P/2014/217
Record Dates: First submitted 2016-09-01; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Implantable Defibrillator User
Keywords: implantable cardioverter defibrillator; primary prevention; psychological follow-up; anxiety; depression; quality of life
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychological follow-up (Experimental): Patients undergoing implantation of an ICD for primary prevention will have an individual interview with a qualified psychologist in addition to standard medical follow-up.
  Interventions: Other: Individual interview with a qualified psychologist
- Control (No Intervention): Patients undergoing implantation of an ICD for primary prevention will have standard medical follow-up.

INTERVENTIONS:
Other: Individual interview with a qualified psychologist — Individual, recorded interview with a qualified psychologist to discuss any and all subjects related to the ICD implantation, or any other topics deemed relevant by the patient.
  Arms: Psychological follow-up

SUMMARY:
This study aims to investigate whether follow-up with a psychologist has an impact on the outcome of patients with an implantable automated defibrillator.

DETAILED DESCRIPTION:
The implantation of an ICD in primary prevention is known to increase the rates of anxiety and depression, which can reach up to 45% and 35% respectively in this patient population. Several studies have reported that psychological accompaniment for these patients can alleviate the symptoms of anxiety and/or depression. Therefore, we aim to investigate the utility of psychological follow-up for a period of 1 year after first implantation of an ICD for primary prevention.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (aged 18 years or over)
* indication for implantation of an ICD for primary prophylaxis
* written informed consent provided
* patients with social security coverage

Exclusion Criteria:

* patients under legal tutorship or guardianship
* patients with no social security coverage
* patients still within the exclusion period after participation in another clinical trial, as indicated by the national registry of clinical trial volunteers
* patients unable to complete the questionnaires (language barriers, mentally deficient, illiteracy or dementia)
* patients awaiting heart transplant
* patients who refuse to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Mini International Neuropsychiatric Interview score | 48 hours after implantation
Mini International Neuropsychiatric Interview score | 2 weeks after implantation
Mini International Neuropsychiatric Interview score | 2 months after implantation
Mini International Neuropsychiatric Interview score | 4 months after implantation
Mini International Neuropsychiatric Interview score | 6 months after implantation
Mini International Neuropsychiatric Interview score | 12 months after implantation

SECONDARY OUTCOMES:
Quality of life | 48 hours after implantation
  Measure of patient's quality of life using the Short Form (SF) 36 item questionnaire
Quality of life | 2 weeks after implantation
  Measure of patient's quality of life using the Short Form (SF) 36 item questionnaire
Quality of life | 2 months after implantation
  Measure of patient's quality of life using the Short Form (SF) 36 item questionnaire
Quality of life | 4 months after implantation
  Measure of patient's quality of life using the Short Form (SF) 36 item questionnaire
Quality of life | 6 months after implantation
  Measure of patient's quality of life using the Short Form (SF) 36 item questionnaire
Quality of life | 12 months after implantation
  Measure of patient's quality of life using the Short Form (SF) 36 item questionnaire
State-Trait Anxiety Inventory | 48 hours after implantation
  Measure of state and trait anxiety
State-Trait Anxiety Inventory | 2 weeks after implantation
  Measure of state and trait anxiety
State-Trait Anxiety Inventory | 2 months after implantation
  Measure of state and trait anxiety
State-Trait Anxiety Inventory | 4 months after implantation
  Measure of state and trait anxiety
State-Trait Anxiety Inventory | 6 months after implantation
  Measure of state and trait anxiety
State-Trait Anxiety Inventory | 12 months after implantation
  Measure of state and trait anxiety
Minnesota Living with Heart Failure questionnaire | 48 hours after implantation
  Evaluation of the quality of life in patients with heart failure
Minnesota Living with Heart Failure questionnaire | 2 weeks after implantation
  Evaluation of the quality of life in patients with heart failure
Minnesota Living with Heart Failure questionnaire | 2 months after implantation
  Evaluation of the quality of life in patients with heart failure
Minnesota Living with Heart Failure questionnaire | 4 months after implantation
  Evaluation of the quality of life in patients with heart failure
Minnesota Living with Heart Failure questionnaire | 6 months after implantation
  Evaluation of the quality of life in patients with heart failure
Minnesota Living with Heart Failure questionnaire | 12 months after implantation
  Evaluation of the quality of life in patients with heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Guignier, MD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Besancon, Besançon, Besancon, France

IPD SHARING:
Plan to Share IPD: No